CLINICAL TRIAL: NCT02386969
Title: Long-term Efficacy of Repetitive Transcranial Magnetic Stimulation on the Primary Motor Cortex (M1) in Central Neuropathic Pain
Brief Title: Repetitive Transcranial Magnetic Stimulation in Central Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1408207; 2015-A00065-44 (Other: ANSM)
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; repetitive transcranial magnetic stimulation (rTMS)
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS then sham rTMS (Experimental): Active rTMS in 1st period and sham rTMS in 2nd period
  Interventions: Device: active rTMS then sham rTMS
- Sham rTMS then active rTMS (Experimental): Sham rTMS in 1st period and active rTMS in 2nd period
  Interventions: Device: sham rTMS then active rTMS

INTERVENTIONS:
Device: active rTMS then sham rTMS — A first period during which the patient will have 1 session of active rTMS every 3 weeks for 3 months A 2nd period during which the patient will have 1 session of sham rTMS every 3 weeks for 3 months
  Arms: Active rTMS then sham rTMS
Device: sham rTMS then active rTMS — A first period during which the patient will have 1 session of sham rTMS every 3 weeks for 3 months A 2nd period during which the patient will have 1 session of active rTMS every 3 weeks for 3 months
  Arms: Sham rTMS then active rTMS

SUMMARY:
The repetitive transcranial magnetic stimulation (rTMS) is used in pain treatment for several years. The aim of the study is to assess, in a rigorous scientific protocol, analgesic effect of the neuronavigated rTMS assisted by robotic arm on chronic neuropathic painful subjects. The crossover study is randomized, double blinded and controlled (sham rTMS) and it includes a large homogeneous population suffering of central neuropathic pain.

DETAILED DESCRIPTION:
The repetitive transcranial magnetic stimulation (rTMS) is used in pain treatment for several years. The latest meta-analysis showed that rTMS has not prove its scientific efficacy. It could be explained by several reasons: poor methodologic quality, stimulations parameters, technologic hardware, ... The aim of the study is to assess, in a rigorous scientific protocol, analgesic effect of the neuronavigated rTMS assisted by robotic arm on chronic neuropathic painful subjects. The crossover study is randomized, double blinded and controlled (sham rTMS) and it includes a large homogeneous population suffering of central neuropathic pain. The stimulated region is the primary motor cortex with high frequency (20Hz). This study has two periods (real and sham) of 12 weeks with four sessions of stimulation per period and 8 weeks of washout between the two.

ELIGIBILITY:
Inclusion Criteria:

* Central neuropathic pain
* Chronic pain with an average pain intensity is greater than or equal to 40/100
* Pain presents a daily or almost daily (at least 4 days out of 7)
* Pain presents for more than 6 months
* Patients who signed informed consent,
* Patients whose pain medication is stable for 15 days before to inclusion, and will not need to be modified for the duration of the study,
* Patients can be monitored for the duration of the study (29 weeks)
* Patients affiliated to a health insurance plan or entitled,
* Patients with a cerebral MRI T1.

Exclusion Criteria:

* Labor dispute or Accident,
* Contraindication to rTMS (treatment with electroconvulsive therapy during the previous month, epilepsy and / or a history of epilepsy, history of head trauma, neurosurgical injury; intracranial hypertension metal clip; pacemaker pregnant or lactating women)
* Abuse of drugs or psychoactive substances
* Peripheral Neuropathic Pain,
* Neuropathic pain within the framework of a progressive disease (HIV, cancer, non-stabilized system disease)
* Intermittent pain,
* Pain in less than 6 months,
* Presence of other pain more severe than that justify inclusion,
* Lack of stability pain scores on two successive evaluations, defined as a change of more than 30% between the two assessments of the average pain between the first two visits (inclusion and first session)
* Patients unable to understand informed consent, under guardianship,
* Patients refusing to stop or can not stop the prohibited treatment during the study,
* Patients participating in another research protocol involving a drug within 30 days before inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Percentage of pain relief (0%= " no pain relief " and 100% " complete pain relief ") | 3 weeks later the last session of rTMS (active ) so week n°12
  Percentage of pain relief compared to the beginning of the period of the study before the first stimulation
Percentage of pain relief (0%= " no pain relief " and 100% " complete pain | 3 weeks later the last session of rTMS (sham) so week n°29.
  Percentage of pain relief compared to the beginning of the period of the study before the first stimulation

SECONDARY OUTCOMES:
Intensity of " average pain " assess by a visual analogue scale (VAS) of 100 mm (0= " no pain " and 100= " worst pain imaginable "). | 3 weeks after the last sessions of rTMS (real or sham), so week n°12 and n°29.
Intensity of " average pain " with VAS before each session compared to the previous meeting (or weeks number: 3, 6, 9, 12 and 20, 23, 26, 29) | before each session (or weeks number: 3, 6, 9, 12 and 20, 23, 26, 29)
Percentage relief of pain before each session compared to the previous meeting (or weeks number: 3, 6, 9, 12 and 20, 23, 26, 29) | before each session (or weeks number: 3, 6, 9, 12 and 20, 23, 26, 29)
Neuropathic dimension | at each session (or weeks number: 0, 3, 6, 9, 12 and 17, 20, 23, 26, 29)
  specific paper questionnaire of neuropathic pain NPSI at each session (or weeks number: 0, 3, 6, 9, 12 and 17, 20, 23, 26, 29)
- Percentage of responders to the treatment real rTMS: subjects whom the Percentage of pain relief at the end of each period of 4 sessions (weeks n°12 and 29) is at least 15%. | at the end of each period of 4 sessions (weeks n°12 and 29)
Consumption of analgesic treatment | 3 weeks before the first session of the period and week : 3, 6, 9, 12 and 20, 23, 26, 29

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France